CLINICAL TRIAL: NCT04388111
Title: Intraosseous Morphine Administration During Primary Total Knee Arthroplasty: A Randomized Clinical Trial
Brief Title: Intraosseous Morphine in Primary TKA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Kwan Park, MD, Principal Investigator, The Methodist Hospital Research Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro000023481
Record Dates: First submitted 2020-05-11; First posted 2020-05-14 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Knee Disease; Arthritis Knee; Pain, Acute
Keywords: Intraosseous; Total knee arthroplasty; Morphine
MeSH Terms: conditions — Acute Pain | interventions — Morphine

STUDY DESIGN:
Intervention Model Description: Group 1: Receives an intraosseous injection of morphine (mixed with standard antibiotics) during their primary total knee replacement or Group 2: Serves as the control group and only receives an intraosseous injection of antibioitics during their total knee replacement.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Patient, provider, and laboratory technicians are blinded to the patient's study group. Only the research coordinator and necessary OR support staff are aware of the patient's study group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control Group (No Intervention): Patient receives an intraosseous injection of antibiotics into the tibia as per the standard of care for primary total knee arthroplasty under the study providers.
- Intarosseous Morphine (Experimental): Patient receives an intraosseous injection of antibiotics + 10mg of morphine into the tibia during their total knee arthroplasty.
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Morphine — 10mg of Morphine delivered Intraosseously
  Arms: Intarosseous Morphine

SUMMARY:
The research team wants to investigate if an intraosseous injection (directly into the bone marrow) of morphine during primary total knee replacement helps with post-operative pain following primary total knee replacement surgery. For this study patients will either be randomized into one of two groups: Group 1: Receives an intraosseous injection of morphine (mixed with standard antibiotics) during their primary total knee replacement or Group 2: Serves as the control group and only receives an intraosseous injection of antibioitics during their total knee replacement. The research team will have patients fill out a symptom journal for two weeks following their surgery to measure pain levels and pain medication consumed throughout the day as well as nausea and other symptoms. Additionally, the research team will take blood samples both intraoperatively and post-operatively (10 hours post-op) to measure the level of inflammatory markers as well as morphine.

ELIGIBILITY:
Inclusion Criteria:

* Patient gives informed consent to participate in the study
* Patient is undergoing a primary total knee arthroplasty.
* Age > 18 and <80 years old.

Exclusion Criteria:

* Patient lacks the capacity to consent to the research project (study will not utilize LAR signatures during the informed consent process)
* Weigh < 100 pounds
* BMI > 35
* Pregnancy or suspected pregnancy
* Past medical history of opioid addiction.
* Established hypersensitivity (ie allergy) to morphine.
* Acute or chronic liver disease for example cirrhosis.
* Use of any narcotics 5 days before surgery (opioids, hydrocodone, morphine, hydromorphone, fentanyl, etc).
* Undergoing bilateral total knee replacement, revision total knee arthroplasty, or any additional procedure outside of a primary total knee arthroplasty.
* Unable to get general and spinal anesthesia.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2020-05-05 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-05-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Houston Methodist Hospital, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited at hospital from 5/5/2020 through 4/1/2021
Period: Overall Study
Arm/Group | Control Group | Intarosseous Morphine
Started | 33 | 32
Completed | 24 | 24
Not Completed | 9 | 8
Not completed — Lost to Follow-up | 5 | 3
Not completed — Adverse Event | 1 | 1
Not completed — Protocol Violation | 2 | 4
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Intarosseous Morphine | Total
Number analyzed (Participants) | 24 | 24 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.06 (6.37) | 65.20 (8.01) | 65.13 (7.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 15 | 26
  Male | 13 | 9 | 22
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24 | 24 | 48
Weight (kg) [Mean (Standard Deviation); unit: KG] | 96.03 (21.74) | 88.13 (15.99) | 92.08 (19.29)
BMI [Mean (Standard Deviation); unit: KG/m^2] | 30.58 (3.89) | 31.36 (5.09) | 30.97 (4.50)

OUTCOME MEASURES:

1. Primary Outcome: Post-operative Pain
Description: Patient will fill out Visual Analog Scale pain scores three times a day for 14 days (day 1 as day of surgery) post-op in a pain journal. Levels will be compared between study groups. A higher score indicates a higher self-perceived level of pain and a lower score indicates a lower perceived level of pain for the patient. "0" representing no pain at all on the scale and "10" representing the highest pain imaginable. Scores are reported 3 times a day per day and averaged for that day. All of these scores were then averaged for the 14 day period and reported below.
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: visual analog pain scale
Arm/Group | Control Group | Intarosseous Morphine
Number analyzed (Participants) | 24 | 24
visual analog pain scale | 4.29 (0.39) | 3.57 (0.37)

2. Secondary Outcome: Knee Injury and Osteoarthritis Outcome Score for Joint Replacement (KOOS Jr) Score - Pre-operative
Description: KOOS Jr Score patient reported outcome measure. Scale is from 0 to 100 with a 0 being total knee disability and 100 being perfect knee health.
Time Frame: preoperative
Measure: Mean (Standard Error); unit: KOOS Jr. Score
Arm/Group | Control Group | Intarosseous Morphine
Number analyzed (Participants) | 24 | 24
KOOS Jr. Score | 52.0 (2.0) | 51.4 (2.1)

3. Secondary Outcome: Knee Injury and Osteoarthritis Outcome Score for Joint Replacement (KOOS Jr) Score - Two Weeks Postoperative
Description: KOOS Jr Score patient reported outcome measure. Scale is from 0 to 100 with a 0 being total knee disability and 100 being perfect knee health. Reported two-weeks post-operative.
Time Frame: two week postoperatively
Measure: Mean (Standard Error); unit: KOOS Jr. Score
Arm/Group | Control Group | Intarosseous Morphine
Number analyzed (Participants) | 24 | 24
KOOS Jr. Score | 57.1 (2.0) | 62.2 (2.1)

4. Secondary Outcome: Knee Injury and Osteoarthritis Outcome Score for Joint Replacement (KOOS Jr) Score - Two Weeks Postoperative
Description: KOOS Jr Score patient reported outcome measure. Scale is from 0 to 100 with a 0 being total knee disability and 100 being perfect knee health. Reported 8 weeks post-operative.
Time Frame: 8 weeks postoperatively
Measure: Mean (Standard Error); unit: KOOS Jr. Score
Arm/Group | Control Group | Intarosseous Morphine
Number analyzed (Participants) | 24 | 24
KOOS Jr. Score | 64.0 (2.2) | 71.5 (2.3)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Control Group | Intarosseous Morphine
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 1/24 | 1/24
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group (N=24) | Intarosseous Morphine (N=24)
Pulmonary Embolism (Blood and lymphatic system disorders) | 1 (1) | 1 (1) — Both groups had a single occurrence of pulmonary embolism in them (each occurred within two weeks of their procedure). This was determined to not be related to the study intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-12): https://cdn.clinicaltrials.gov/large-docs/11/NCT04388111/Prot_SAP_000.pdf